CLINICAL TRIAL: NCT02073669
Title: Better Identification of Latent Tuberculosis Infection Among Israeli Young Adults by Comparison Skin Tests and Interferon Gamma Releasing Assays (IGRA)
Brief Title: Latent Tuberculosis in Second Generation Immigrants From High Risk Countries Compare to Low-risk Young Israeli Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel Aviv Lung Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SHEBA-13-0668-DS-CTIL
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Latent Tuberculosis
Keywords: latent tuberculosis; tuberculin skin test; Interferon gamma release assay; immigration
MeSH Terms: conditions — Latent Tuberculosis | interventions — Blood Specimen Collection; Interferon-gamma Release Tests

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Second generation immigrants from high TB incidence countries (Other): Answering the study Questionnaire and blood sampling for Interferon gamma release assay (IGRA).
  Interventions: Procedure: Answering the study Questionnaire and blood sampling for Interferon gamma release assay (IGRA)
- Native Israelis (Other): Answering the study Questionnaire and blood sampling for Interferon gamma release assay (IGRA).
  Interventions: Procedure: Answering the study Questionnaire and blood sampling for Interferon gamma release assay (IGRA)

INTERVENTIONS:
Procedure: Answering the study Questionnaire and blood sampling for Interferon gamma release assay (IGRA)

SUMMARY:
The aim of study is to evaluate the prevalence of latent TB in second generation immigrants from countries with high incidence of tuberculosis (above 20 of 100,000) compare to the control native Israelis without a family member who was born in a country with high incidence of tuberculosis. Using study questionnaire IGRA and tuberculin skin test the investigators expect that the second generation immigrants group will have more positive IGRA test than the control native group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25
* Men and women
* Second generation immigrants from countries with high incidence of tuberculosis (above 20 of 100,000).
* Native Israelis without a family member who was born in a country with high incidence of tuberculosis.

Exclusion Criteria:

* Prior contact with a tuberculosis patient
* Working (more than a month) in high risk setting such as health care workers, working with immigrants from countries with high incidence of tuberculosis.
* HIV infection and any immunodeficiency condition.
* Recent live-virus vaccination
* Acute infectious disease
* Prior serious reaction to tuberculin skin test
* Pregnancy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Interferon gamma release assay ( IGRA) | Up to 3 months after tuberculin skin test

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Sheba Medical Center, Ramat Gan
  - Israeli Defense Forces, Ramat Gan